CLINICAL TRIAL: NCT05606692
Title: Impact of Propofol-Based Total Intravenous Anesthesia Versus Anesthesia With Sevoflurane on Long-term Outcomes With Patients Undergoing Elective Surgery for Primary Ovarian Cancer
Brief Title: Influences of Propofol and Sevoflurane Anesthesia in Ovarian Cancer (Anesthetics)
Acronym: anesthetics
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20220157
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Cancer
Keywords: Primary Ovarian Cancer; Propofol; Sevoflurane; Survival
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane group (Active Comparator): The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3).
  Interventions: Drug: Sevoflurane/Ultane
- Propofol group (Experimental): The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Interventions: Drug: Propofol 1%

INTERVENTIONS:
Drug: Propofol 1% — The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Other Names: ANESVAN INJECTION 10MG/ML (PROPOFOL) "CHI SHENG"
  Arms: Propofol group
Drug: Sevoflurane/Ultane — The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3).
  Other Names: Sevoflurane/ Ultane 250mL/Bot
  Arms: Sevoflurane group

SUMMARY:
Ⅶ. Study procedures (summary)

1. Written informed consent must be obtained before any study specific procedures are undertaken.

   Qualified participants were identified at the pre-anesthesia evaluation clinic or ward. The informed consents are obtained from the patient in the ward at night before the operation.
2. The process of the experiment (brief describe) In the preoperative waiting area, the patients are randomly assigned and divided into two groups according to the allocation sequence table (corresponding to 1:1 randomization) generated by the computer. The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system. The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3). During the operation, the dose of anesthetic drugs (propofol/fentanyl /remifentanil and sevoflurane/cisatracurium/rocuronium) are adjusted to maintain the mean arterial pressure and heartbeat fluctuations within 20% of the baseline value and Entropy (or BIS) value at 40-60in both groups. The following patient data were recorded, the type of anesthesia, sex, age at the time of surgery, preoperative Karnofsky performance status (KPS) score and functional capacity, the postoperative complications within 30 days (according Clavien-Dindo classification), ASA physical status scores, tumor marker ,tumor size, intraoperative blood loss/transfusion, duration of surgery, duration of anesthesia, total opioid (remifentanil/fentanyl) use, postoperative radiation therapy, postoperative chemotherapy, postoperative concurrent chemoradiotherapy, the presence of disease progression, and 6-month, 1-year, 3-year and 5-year overall survival and Karnofsky performance status score were recorded.

DETAILED DESCRIPTION:
During the operation, the dose of anesthetic drugs (propofol/ fentanyl /remifentanil and sevoflurane/ cisatracurium/ rocuronium) are adjusted to maintain the mean arterial pressure and heartbeat fluctuations within 20% of the baseline value and Entropy (or BIS) value at 40-60in both groups. The following patient data were recorded, the type of anesthesia, age at the time of surgery, preoperative Karnofsky performance status (KPS) score and functional capacity, the postoperative complications within 30 days (according Clavien-Dindo classification), ASA physical status scoress, tumor marker , tumor size, intraoperative blood loss/transfusion, duration of surgery, duration of anesthesia, total opioid (remifentanil/ fentanyl/ propofol) use, postoperative radiation therapy, postoperative chemotherapy, postoperative concurrent chemoradiotherapy, the presence of disease progression, and 6-month, 1-year, and 3-year overall survival and Karnofsky performance status score were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Twenty to eighty-year-old.
2. ASA class I-III.
3. Patients undergoing elective craniotomy for primary ovarian tumors under general anesthesia.

Exclusion Criteria:

1. Severe mental disorder
2. Poor liver function
3. Pregnant or lactating women
4. Morbid obesity
5. Have a history of allergy to any drug used in this study
6. Non-primary ovarian cancer surgery
7. Undergoing ovarian cancer pathological section surgery
8. Patients with incomplete medical records
9. Combined with other surgeries, emergency surgeries
10. Concomitant patients with other non-ovarian cancer therapy
11. Patients receiving palliative treatment after ovarian cancer surgery
12. During the maintenance period of anesthesia, propofol or sevoflurane should not be used as anesthetic drugs
13. Intraoperative combined use of multiple anesthetics (such as ketamine, dexmedetomidine, other inhalation anesthetics)
14. Those diagnosed with benign tumors before and after surgery
15. Patients with metastases to the ovary

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5 years
  progression-free survival

SECONDARY OUTCOMES:
6-month overall survival | 6 months
  6-month overall survival
1-year overall survival | 1 year
  1-year overall survival
3-year overall survival | 3 years
  3-year overall survival
5-year overall survival | 5 years
  5-year overall survival
Karnofsky performance score | 5 years
  Karnofsky performance score, from 100 to 0, where 100 is perfect health and 0 is death. The lower the Karnofsky performance score, the worse the likelihood of survival.
postoperative complications | 30 days
  postoperative complications within 30 days (according Clavien-Dindo classification)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Fu Wu, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan